CLINICAL TRIAL: NCT01461928
Title: A Randomized Study Comparing Maintenance Therapy With Subcutaneous Rituximab Continued Until Progression With Observation Only in Patients With Relapsed or Refractory, Indolent Non-Hodgkin's Lymphoma Who Completed and Responded to Rituximab-based Immunochemotherapy Induction and Initial 2-year Rituximab Maintenance Therapy Administered Subcutaneously
Brief Title: A Study Comparing Maintenance Subcutaneous Rituximab With Observation Only in Participants With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma Who Had Responded to Rituximab-based Immunochemotherapy Induction and 2-year Maintenance With Subcutaneous Rituximab
Acronym: MabCute
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO25455; 2010-023407-95 (EudraCT Number)
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Maintenance II Period Observation Only (Other): Participants will receive standard chemotherapy regimen in combination with 375 mg/m^2 rituximab IV in Cycle 1 (3-4 week-cycles), followed by 1400 mg rituximab SC every 3-4 weeks for 8 cycles (induction period); 1400 mg rituximab SC every 8 weeks for 24 months (Maintenance I period); no treatment in Maintenance II period until disease progression or end of study, whichever occurs first.
  Interventions: Drug: Chemotherapy (Induction Period); Drug: Rituximab
- Maintenance II Period Rituximab (Experimental): Participants will receive standard chemotherapy regimen in combination with 375 mg/m^2 rituximab IV in Cycle 1 (3-4 week-cycles), followed by 1400 mg rituximab SC every 3-4 weeks for 8 cycles (induction period); 1400 mg rituximab SC every 8 weeks for 24 months (Maintenance I period); 1400 mg rituximab SC every 8 weeks until disease progression or end of study, whichever occurs first (Maintenance II period).
  Interventions: Drug: Chemotherapy (Induction Period); Drug: Rituximab

INTERVENTIONS:
Drug: Chemotherapy (Induction Period) — Participants will receive standard combination chemotherapy every 3-4 weeks for 6 to 8 months. The chemotherapy regimen will be selected at Investigator's discretion, for individual participant. Study protocol does not enforce any particular chemotherapy regimen.
Drug: Rituximab — Participants will receive rituximab according to the regimen specified in individual arm.
  Other Names: Rituxan; MabThera; RO0452294

SUMMARY:
This multicenter, randomized, open-label, parallel-group study will evaluate the efficacy and safety of subcutaneously administered rituximab in comparison with observation only as maintenance therapy in participants with relapsed or refractory indolent Non-Hodgkin's lymphoma (NHL). All participants will receive induction therapy with rituximab (375 milligrams per square meter [mg/m^2] intravenously [IV] in Cycle 1, then 1400 mg subcutaneous [SC] every 3-4 weeks) plus standard chemotherapy for 6-8 months; followed by 24 months of maintenance I period with rituximab (1400 mg SC every 8 weeks). Participants completing therapy and showing partial or complete response will be randomized to receive either rituximab (1400 mg SC every 8 weeks) or observation with no treatment during maintenance II period and will be followed for at least 15 months. Anticipated time on study treatment is until disease progression, unacceptable toxicity or end of study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Cluster of Differentiation 20-positive (CD20+) follicular NHL Grade 1, 2 or 3a, or other CD20+ indolent NHL (Waldenström's macroglobulinemia or lymphoplasmacytic lymphoma, marginal zone lymphoma) according to World Health Organization (WHO) classification system
* Participants must have received and must have relapsed or been refractory to, one or more lines of adequate therapy prior to enrollment, including at least one line consisting of immunotherapy and/or chemotherapy and/or radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2

Exclusion Criteria:

* Transformation to high-grade lymphoma
* Aggressive lymphoma (for example, mantle cell lymphoma [MCL])
* Presence or history of central nervous system (CNS) lymphomatous disease
* Other malignancy within 5 years prior to enrollment, except for curatively treated carcinoma in situ of the cervix, squamous cell carcinoma of the skin or basal cell skin cancer, or cervical carcinoma Stage 1B or less, breast cancer in situ or localized prostate cancer Stage T1c if treated with curative intent and relapse- and metastasis-free for at least 2 years prior to enrollment
* Inadequate hematological, hepatic or renal function
* Known human immunodeficiency virus (HIV) infection
* Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B or C)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (180):
- University "Mother Theresa" Hospital Center; Oncology Department, Tirana, Albania
- Argentina (3):
  - CEMIC Saavedra, Buenos Aires
  - Instituto Damic, Córdoba
  - Hospital Privado de Comunidad; Oncology, Mar del Plata
- Austria (5):
  - Lkh-Univ. Klinikum Graz; Klin. Abt. Für Hämatologie, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Innere Medizin Abt. Für Hämatologie & Onkologie, Innsbruck
  - Kepler Universitätskliniken GmbH - Med Campus III; III. Medizinische Abteilung, Linz
  - Landeskrankenhaus Rankweil; Interne E, Rankweil
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Hämatologie & Hämostaseologie, Vienna
- Brazil (8):
  - Centro de Tratamento Oncologico - CETRON, Rio de Janeiro, Rio de Janeiro
  - Hospital da Cidade de Passo Fundo; Centro de Pesquisa em Oncologia, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP; Hematologia, São Paulo, São Paulo
  - Hospital Santa Marcelina;Oncologia, São Paulo, São Paulo
- Bulgaria (3):
  - UMHAT Dr Georgi Stranski; Hematology, Pleven
  - Tokuda Hospital Sofia; Hematology department, Sofia
  - UMHAT Alexandrovska EAD; Hematology, Sofia
- Colombia (3):
  - Centro Javeriano de Oncología, Bogotá
  - Fundacion Santa Fe de Bogotá, Bogotá
  - Instituto Nacional de Cancerologia; Hematology, Bogotá
- Ecuador (4):
  - Hospital Abel Gilbert Ponton; Oncology, Guayaquil
  - Teodoro Maldonado Carbo Hospital; Oncology Service, Guayaquil
  - Hospital Solca Portoviejo; Oncologia, Portoviejo
  - Hospital Solca Quito; Oncologia, Quito
- Kasr Eieny Uni Hospital; Oncology (Nemrock), Cairo, Egypt
- France (26):
  - Centre Hospitalier Uni Ire; Service Des Maladies Du Sang, Angers
  - CH Henri Mondor; Med Interne Neuro Endocrinologie, Aurillac
  - Centre Hospitalier de La Cote Basque; Hematologie, Bayonne
  - Hopital Jean Minjoz; Hematologie, Besançon
  - Hopital Augustin Morvan; Hematologie, Brest
  - Institut d'Hématologie de Basse Normandie, Caen
  - CH Metropole de Savoie, Chambéry
  - Chu Estaing; Hematologie Clinique Adultes, Clermont-Ferrand
  - Ch Sud Francilien; Hematologie Oncologie, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - Chu Site Du Bocage;Hematologie Clinique, Dijon
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Hôpital Albert Michallon; Hematologie Clinique, La Tronche
  - Hopital Andre Mignot; Hematologie - Oncologie, Le Chesnay
  - Ch Du Mans; Medecine Hematologie Oncologie, Le Mans
  - Hopital Claude Huriez; Hematologie, Lille
  - Hopital Uni Ire Dupuytren; Hematologie, Limoges
  - Hopital Nord; Laboratoire D'Hematologie, Marseille
  - Hôpital Lapeyronie; Hématologie Oncologie Médicale, Montpellier
  - Hopital Emile Muller; Hematologie, Mulhouse
  - Hopital Hotel Dieu Et Hme; Clinique Dermatologique, Nantes
  - Centre Antoine Lacassagne;B4 Hematologie Cancerologie, Nice
  - Hopital Pitie Salpetriere; Hematologie Clinique, Paris
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
  - Centre Henri Becquerel; Hematologie, Rouen
  - Hopital Purpan; Hematologie Clinique, Toulouse
- Germany (25):
  - Gemeinschaftspraxis Dr. Bueckner und Dr. Nueckel, Bochum
  - Klinikum Darmstadt GmbH; Med. Klinik V; Onkologie & Hämatologie, Darmstadt
  - St. Johannes Hospital; Abt. für Hämatologie und Onkologie, Dortmund
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Gemeinschaftspraxis Dr. med. J. Mohm und Dr. med. G. Prange-Krex; Fachaerzte fuer Innere Medizin, Dresden
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Internistisch-Onkologische Gemeinschaftspraxis; Dres. Rohrberg, Hurtz, Schma usw., Halle
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Onkologische Schwerpunktpraxis (Eps-Gmbh), Jena
  - Dres. Richard Hansen Susanne Pfitzner-Dempfle und Manfred Reeb, Kaiserslautern
  - Dres. Barbara Tschechne Stefanie Luft und Wolf-Oliver Jordan, Lehrte
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Gemeinschaftspraxis Fr. Dr. med. Balser & Hr. Dr. med. Weidenbach, Marburg
  - Dres. Michael Maasberg Marion Schmitz und Maria Theresia Keller, Mayen
  - Staedtisches Krankenhaus Muenchen-Schwabing, Haematologie & Onkolgie, München
  - Hamatol Onkol Praxisgemeinschaft Dres H H-D Schick/D Schick, München
  - Klinikum Grosshadern der LMU, München
  - Klinikum rechts der Isar der TU München; III. Medizinischen Klinik (Hämatologie/Onkologie), München
  - Praxis Dr.med. Jens Uhlig, Naunhof
  - Oncologianova GmbH, Recklinghausen
  - Klinik der Uni Regensburg; Hämatologie/Onkologie, Studienzentrale, Regensburg
  - Dres. Andreas Hübner, Andreas Lück und Petra Bruhn, Rostock
  - Dres. Ulrich Banhardt und Thomas Fietz, Singen
  - Dres. Emil Höring Matthias Respondek und Ulrike Schwinger, Stuttgart
- Greece (5):
  - General Hospital of Athens Evangelismos; Hematology, Athens
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - University Hospital of Ioannina; Hematology, Ioannina
  - University Hospital of Larissa; Hematology Dept., Larissa
  - University Hospital Of Patras; Dept. Of Internal Medicine-Hematology Division, Pátrai
- Hungary (5):
  - Semmelweis University, First Dept of Medicine, Budapest
  - St Laszlo Hospital, Pharmacy, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - Uni of Debrecen; 2Nd Clinic of Internal Medicine, Debrecen
  - University of Pecs, I st Dept of Internal Medicine, Pécs
- Italy (20):
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - A.O. Universitaria Federico II Di Napoli; Oncologia Ed Endocrinologia Clinica, Napoli, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - A.O.U. Policlinico di Modena-Dipartimento di Medicina Diagnostica, Clinica e di Sanità pubblica, Modena, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Ematologica, Udine, Friuli Venezia Giulia
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova; Ematologia 1, Genoa, Liguria
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - Azienda Sanitaria Di Bolzano; Ematologia E Centro Trapianto Mid.Osseo, Bolzano, Trentino-Alto Adige
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
  - A.O. Universitaria Senese; Ematologia, Siena, Tuscany
  - Uni Degli Studi; Dip.Med.Clinica E Sperim. Ematologia, Padua, Veneto
  - Ospedale Ca Foncello; Ematologia, Treviso, Veneto
  - Uni Di Verona Policlinico G.B. Rossi; Divisione E Cattedra Di Ematologia, Verona, Veneto
- Seamen' Hospital' Dept. of haematology, Klaipėda, Lithuania
- Norway (4):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF; Radiumhospitalet, Oslo
  - Helse Stavanger HF, Stavanger Universitetssjukehus; Klinikk for Blod og kreftsykdommer, Stavanger
  - St. Olavs Hospital HF, Kreftavdelingen, Gastrosentret, Trondheim
- Romania (6):
  - Policlinica de Diagnostic Rapid, Brasov
  - County Clinical Emergency Hospital Brasov, Brasov
  - Institutul Clinic Fundeni; Hematologie, Bucharest
  - Spitalul Clinic Coltea; Clinica de Hematologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu-Mures; compartiment Hematologie, Târgu Mureş
  - Spitalul Clinic municipal de Urgenta Timisoara; Clinica de Hematologie, Timișoara
- Russia (8):
  - Regional Oncology Center, Chelyabinsk
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - Rus Med Academy for Postgraduate Education; Oncology Department, Moscow
  - City Clin Hosp n.a. S.P.Botkin, Moscow
  - Regional Clinical Hospital N.A. Semashko; Hematology, Nizhny Novgorod
  - SRI of Hematology and Transfusiology, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Petrov Research Inst. of Oncology, Saint Petersburg
- Slovakia (2):
  - National Oncology Inst. ; Dept. of Haematology, Bratislava
  - Uni Hospital ; Dept. of Haematol. & Transfusion Medicine, Martin
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (20):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Hematologia, Badalona, Barcelona
  - Hospital de Jerez de la Frontera; Servicio de Hematologia, Jerez de la Frontera, Cadiz
  - Hospital Quiron de Madrid; Servicio de Hematologia, Pozuelo de Alarcón, Madrid
  - Hospital Univ. Central de Asturias; servicio de Hematologia, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias;servicio de Hematologia, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de la Santa Creu i Sant Pau; Servicio de Hematologia, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Hematologia, Cáceres
  - Hospital Universitario San Cecilio; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen- Hospital Universitario Medico Quirurgico; Servicio de Hematologia, Jaén
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio Hematologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Hematologia, Málaga
  - Complejo Hospitalario Universitario de Ourense, Servicio de Hematologia, Ourense
  - Hospital Arnau de Vilanova (Valencia) Servicio de Hematologia, Valencia
  - Complejo Hospitalario Zamora- H. Virgen de la Concha; Servicio de Hematología, Zamora
  - Hospital Royo Villanova; Servicio de Hematologia, Zaragoza
- Sweden (6):
  - Laenssjukhuset; Medicinkliniken/Hematologsektionen, Halmstad
  - Sunderby Sjukhus; Medicinkliniken, Luleå
  - Capio, S:T Gorans Hospital; Dept of Medicine, Stockholm
  - Södersjukhuset, Medicinkliniken/Sektionen för Hematologi, Stockholm
  - Uddevalla Sjukhus; Medicinkliniken, Uddevalla
  - Västmanlands sjukhus Västerås, Onkologmottagningen, Västerås
- Switzerland (2):
  - Ospedale San Giovanni; Oncologia, Bellinzona
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich
- Turkey (Türkiye) (6):
  - GATA (Gulhane Military Medical School), Ankara
  - Hacettepe Uni Medical Faculty; Hematology, Ankara
  - Gazi Uni Medical School; Hematology, Ankara
  - Istanbul Uni Capa Medical Faculty; Inst. of Oncology, Istanbul
  - Marmara University Pendik Training and Research Hospital, Hematology Department, Istanbul
  - Erciyes Uni ; Hematology, Kayseri
- United Kingdom (15):
  - Birmingham Heartlands Hospital; Department of Haematology, Birmingham
  - Royal Bournemouth General Hospital; Haematology, Bournemouth
  - Addenbrookes Hospital; Haematology, Cambridge
  - Kent & Canterbury Hospital; Clinical Haematology, Canterbury
  - Uni Hospital of Wales; Dept of Haematology, Cardiff
  - Leicester Royal Infirmary; Dept of Haematology, Leicester
  - Royal Liverpool Uni Hospital; Haematology, Liverpool
  - University College London, Department of Haematology, London
  - The Royal Marsden Hospital; Dept of Medicine, London
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk & Norwich Hospital; Dept of Haematology, Norwich
  - Nottingham City Hospital; Dept of Haematology, Nottingham
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Derriford Hospital; Haematology, Plymouth
  - Royal Marsden Hospital; Dept. of Medicine, Sutton

REFERENCES:
- [Derived] Rule S, Barreto WG, Briones J, Carella AM, Casasnovas O, Pocock C, Wendtner CM, Zaja F, Robson S, MacGregor L, Tschopp RR, Nick S, Dreyling M. Efficacy and safety assessment of prolonged maintenance with subcutaneous rituximab in patients with relapsed or refractory indolent non-Hodgkin lymphoma: results of the phase III MabCute study. Haematologica. 2022 Feb 1;107(2):500-509. doi: 10.3324/haematol.2020.274803. PMID 34134469
- [Derived] Theodore-Oklota C, Humphrey L, Wiesner C, Schnetzler G, Hudgens S, Campbell A. Validation of a treatment satisfaction questionnaire in non-Hodgkin lymphoma: assessing the change from intravenous to subcutaneous administration of rituximab. Patient Prefer Adherence. 2016 Sep 13;10:1767-1776. doi: 10.2147/PPA.S108489. eCollection 2016. PMID 27695295
- [Derived] Rule S, Collins GP, Samanta K. Subcutaneous vs intravenous rituximab in patients with non-Hodgkin lymphoma: a time and motion study in the United Kingdom. J Med Econ. 2014 Jul;17(7):459-68. doi: 10.3111/13696998.2014.914033. Epub 2014 May 7. PMID 24720836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified for potential recruitment using pre-screening enrolment logs.
Pre-assignment Details: Participants were treated with an induction regimen (6 months) and received SC rituximab at a dose of 375 mg/m2 with chemotherapy followed by 2 years of Maintenance I SC rituximab of 1400 mg alone. Responding participants at the end of Maintenance I were randomized to either Maintenance II rituximab treatment or observation only.
Groups:
- All Participants: Participants were enrolled in an Induction period (up to 8 months) and received SC rituximab at a dose of 375 mg/m2 body surface area (BSA) followed by standard chemotherapy then continued into Maintenance I period (up to 24 months) and received SC rituximab of 1400 mg without chemotherapy. Participants who completed the Induction and Maintenance I periods with SC rituximab and for whom Partial Response (PR) or Complete Response (CR) was confirmed, were considered responders and were then randomized to receive either prolonged SC rituximab continued until disease progression or until the end of study (Maintenance II; Rituximab arm) or observation with no further treatment until the end of study (Maintenance II; Observation arm).
- Maintenance II - Arm A (Rituximab): Participants were randomized to receive SC rituximab administered as a single injection of 1400 mg fixed dose without chemotherapy every 8 weeks until disease progression or until the end of study.
- Maintenance II - Arm B (Observation Only): Participants were randomized to no longer receive SC rituximab but observed until the end of study.
Period: Induction (up to 8 Months)
Arm/Group | All Participants | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only)
Started (Induction period only) | 692 | 0 | 0
Completed (Induction period only) | 494 | 0 | 0
Not Completed | 198 | 0 | 0
Not completed — Adverse Event | 76 | 0 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Physician Decision | 9 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 0 | 0
Not completed — Disease progression | 45 | 0 | 0
Not completed — Eligibility criteria deviation | 10 | 0 | 0
Not completed — Completed Induction, no Maint I received | 11 | 0 | 0
Not completed — Not responding to treatment | 11 | 0 | 0
Not completed — Termination of study in Switzerland | 1 | 0 | 0
Not completed — Treated before eligibility was confirmed | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 0 | 0
Not completed — Protocol deviation | 2 | 0 | 0
Not completed — Prednisolone given prior to enrolment | 1 | 0 | 0
Not completed — Cycle 7 rituximab not given in error | 1 | 0 | 0
Not completed — Promotor request | 1 | 0 | 0
Not completed — Exceeded time limit for next cycle | 1 | 0 | 0
Not completed — Medical advisor request | 1 | 0 | 0
Period: Maintenance I (24 Months)
Arm/Group | All Participants | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only)
Started (Maintenance I only) | 494 | 0 | 0
Completed (Maintenance I only) | 276 (Responders during 2 yrs Maint I treatment) | 0 | 0
Not Completed | 218 | 0 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Diseases progression | 91 | 0 | 0
Not completed — Adverse Event | 70 | 0 | 0
Not completed — Physician Decision | 9 | 0 | 0
Not completed — Did not meet randomization criteria | 2 | 0 | 0
Not completed — Did not perform scheduled assessment | 2 | 0 | 0
Not completed — Delay in rituximab administration | 1 | 0 | 0
Not completed — Not compliant | 1 | 0 | 0
Not completed — Did not meet criteria | 5 | 0 | 0
Period: Maintenance II (15 Months)
Arm/Group | All Participants | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only)
Started (Maintenance II only) | 0 | 138 | 138
Completed (Maintenance II only) | 0 | 115 (6 participants did not receive treatment) | 111
Not Completed | 0 | 23 | 27
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Death | 0 | 10 | 8
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Moved to another town | 0 | 1 | 0
Not completed — Disease progression | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 9 | 8
Not completed — Changed physician in another hospital | 0 | 0 | 1
Not completed — Squamous lung carcinoma | 0 | 0 | 1
Not completed — Withdrew informed consent | 0 | 0 | 1
Not completed — Refused to be transferred to other site | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was used for the analysis of secondary efficacy parameters and Baseline variables. The randomised ITT population (ITTrand) included only randomised participants of Maintenance II period and was used for the analysis of the primary efficacy endpoint of PFS and the secondary analysis endpoint overall survival (OS)
Arm/Group | All Participants
Number analyzed (Participants) | 692
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 346
  Male | 346
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 579
  Black | 7
  Asian | 5
  Other | 32
  Not applicable as per local regulation | 69

OUTCOME MEASURES:

1. Primary Outcome: Maintenance II: Progression-free Survival (PFS) Using 1999 International Working Group (Cheson) Response Criteria for Lymphoma or by the Recommendations for Waldenström's Macroglobulinemia
Description: Progression free survival from randomization (PFSrand) is defined as the time from date of randomization to the date of first documented disease progression or death, whichever occurs first. One participant died in Induction before randomization and one participant died in Maintenance II Observation arm due to an SAE and were not considered in the analysis as no death page was completed. The Observation arm did not include one participant with AE outcome of death reported retrospectively 2 months after discontinuation from study (censored as having no event on Day 456 post-randomization).
Time Frame: From randomization (Maintenance II) up to disease progression or death, whichever occurs first (up to approximately 24 months)
Population: The primary efficacy analysis population was the ITT population (ITTrand), which included only randomised participants (Maintenance II only) and was used for the analysis of the primary efficacy endpoint of PFS and the secondary analysis endpoint overall survival (OS). The PFS end point was not reached.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only)
Number analyzed (Participants) | 138 | 138
Months | NA [NA to NA] — The endpoint could not be analyzed due to the limited number of PFS events | NA [39.75 to NA] — The endpoint could not be analyzed due to the limited number of PFS events
Statistical Analysis 1: Comparison: Maintenance II - Arm A (Rituximab) vs Maintenance II - Arm B (Observation Only); The stratified log rank test p-value was derived using the following randomization stratification strata : Follicular Lymphoma International Prognostic Index (FLIPI) risk category (low, intermediate, high) and indolent NHL subtype (follicular lymphoma, non-follicular lymphoma). Power at time of final analysis was less than 40%. Final analysis was not able to address it's primary objective; Test type: Superiority; p = 0.410, Stratified Long-rank — Power at time of final analysis was less than 40%. Final analysis was not able to address its primary objective; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.37 to 1.53]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, and Infusion/Administration-related Reactions (IRRs/ARRs)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Not all AEs were followed up for the randomized Observation arm. Only Serious AEs and AE grade 3-5 (obtained retrospectively) were collected for this arm. Therefore arms are not comparable overall.
Time Frame: From day of first rituximab induction dose up to day of disease progression, or discontinuation of treatment for any reason (up to approximately 87 months)
Population: The safety population included all participants who received at least one dose of study drug and had a safety assessment performed post randomization.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 692
Participants
  Number of Participants with Adverse Events | 643
  Number of Participants with Serious Adverse Events | 339
  Number of Participants with IRRs/ARRs | 330

3. Secondary Outcome: Event-free Survival (Time to Treatment Failure) Using 1999 International Working Group (Cheson) Response Criteria for Lymphoma or by the Recommendations for Waldenström's Macroglobulinemia
Description: Event-Free Survival was measured from the day of first rituximab Induction dose through Maintenance I and Maintenance II rituximab arm until the date of any treatment failure, including disease progression, or discontinuation of treatment for any reason (e.g. disease progression, toxicity, patient preference, initiation of new anti-lymphoma treatment, or death). Treatment discontinuation was considered as an event and was not applicable to the randomized observation arm.
Time Frame: From day of first rituximab induction dose up to day of any treatment failure, including disease progression, or discontinuation of treatment for any reason (up to approximately 87 months)
Population: All participants who were enrolled into the given study period and had received at least one dose of study treatment at any time were included in the ITT population for each period of the study; Induction, Maintenance I and Maintenance I
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Maintenance II - Arm A (Rituximab) | All Participants
Number analyzed (Participants) | 138 | 692
Months | 65.38 [60.98 to NA] — Not reached because the upper 95% CI of median could not be calculated based on Greenwood formula due to limited events. | 24.99 [20.73 to 27.99]

4. Secondary Outcome: Time to Next Lymphoma Treatment (TNLT)
Description: Time to next lymphoma treatment (TNLT) is defined as the time from date of first rituximab induction dose to the date date of first documented intake of any new antilymphoma treatment (chemotherapy, radiotherapy, immunotherapy, etc.).
Time Frame: From day of first rituximab induction dose up to any new lymphoma treatment (up to approximately 87 months)
Population: The analysis population was the randomised ITT population (ITTrand), which included only randomised participants (Maintenance II only) as well as the ITT population, that included all participants who had completed a Baseline visit and at least one on-treatment assessment (Induction, Maintenance I and Maintenance II).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only) | All Participants
Number analyzed (Participants) | 138 | 138 | 692
Months | NA [NA to NA] — The end point could not be analyzed due to the limited number of events. | NA [NA to NA] — The end point could not be analyzed due to a limited number of events. Biased as subjects stopped treatment and were likely to receive NLT earlier. | NA [NA to NA] — The end point could not be analyzed due to the limited number of events.

5. Secondary Outcome: Overall Survival
Description: Overall survival from first induction treatment (OSRegist) is defined as the time from date of first rituximab induction dose to the date of death, irrespective of cause. One participant died in Induction before randomization and one participant died in Maintenance II Observation arm due to an SAE and were not considered in the analysis as no death page was completed.
Time Frame: From day of first rituximab induction dose up to death (up to approximately 87 months)
Population: The ITT population included all participants who had completed a Baseline visit and at least one on-treatment assessment and were enrolled into each period of the study; Induction, Maintenance I and Maintenance II.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 692
Months | NA [NA to NA] — The end point could not be analyzed due to a limited number of events. Randomized arms pooled as it included information prior to randomization. Interpret with caution.

6. Secondary Outcome: Maintenance II: Overall Survival
Description: Overall survival from randomization (OSrand) is defined as the time from date of randomization to the date of death, irrespective of cause.
Time Frame: From randomization (Maintenance II) up to death (up to approximately 24 months)
Population: The analysis population was the randomised ITT population (ITTrand), which included only randomised participants (Maintenance II only) and was used for the analysis of the primary efficacy endpoint of PFS and the secondary analysis endpoint overall survival (OS).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Maintenance II - Arm A (Rituximab) | Maintenance II - Arm B (Observation Only)
Number analyzed (Participants) | 138 | 138
Months | NA [NA to NA] — The end point could not be analyzed due to the limited number of events | NA [NA to NA] — The end point could not be analyzed due to the limited number of events

7. Secondary Outcome: Percentage of Participants With Partial or Complete Tumor Response (PR/CR) Assessment at End of Induction Using 1999 International Working Group Response Criteria for Lymphoma or by the Recommendations for Waldenström's Macroglobulinemia
Description: Overall response rate is defined as the proportion of responders at the end of the Induction period. A responder is defined as a participant experiencing either CR or PR tumor response according to the Cheson response criteria for indolent lymphoma or the recommendations for Waldenström's macroglobulinemia.
Time Frame: From day of first rituximab induction dose up to end of induction period (up to approximately 8 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 692
Percentage of Participants | 84.7 [81.8 to 87.3]

8. Secondary Outcome: Maintenance I: Percentage of Participants With Conversion of PR to CR Using 1999 International Working Group (Cheson) Response Criteria for Lymphoma or by the Recommendations for Waldenström's Macroglobulinemia
Time Frame: From day of first rituximab induction dose up to end of Maintenance I period (up to approximately 32 months)
Population: The Maintenance I participant analysis group consisted of a subgroup of responding participants who completed Induction and successfully enrolled into Maintenance I. Participants who had partial response (PR) at the end of Induction were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- Maintenance I: Participants received 12 cycles of rituximab administered as a single SC injection of 1400 mg without chemotherapy every 8 weeks for 2 years
Arm/Group | Maintenance I
Number analyzed (Participants) | 357
Percentage | 21.6 [17.4 to 26.2]

9. Secondary Outcome: Progression-free Survival (PFS) Using 1999 International Working Group (Cheson) Response Criteria for Lymphoma or by the Recommendations for Waldenström's Macroglobulinemia
Description: Progression free survival from first induction treatment (PFSregist) is defined as the time from date of first rituximab induction dose to the date of first documented disease progression or death by any cause, whichever occurs first.
Time Frame: From day of first rituximab induction dose up to disease progression or death, whichever occurs first (up to approximately 87 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 692
Months | 59.33 [50.33 to 71.36]

ADVERSE EVENTS:
Time Frame: From Baseline up to 47 months
Description: The SAF population included all participants who had received at least one dose of rituximab during the study (Induction, Maint I, Maint II) and were assigned to treatment groups. Not all AEs were followed up for the randomized Observation arm. Only Serious AEs and AE grade 3-5 were collected for this arm, therefore arms are not comparable overall. All AEs reported in Arm A and Arm B are also included in All Participants.
Groups:
- Arm A: Subjects received SC rituximab administered as a single injection of 1400 mg fixed dose without chemotherapy every 8 weeks until disease progression or until the end of study.
- Arm B (Observation Only): Subjects did not receive further rituximab treatment until the end of study.
Arm/Group | Arm A | Arm B (Observation Only) | All Participants
All-Cause Mortality (participants affected / at risk) | 10/138 | 8/138 | 161/692
Serious Adverse Events (participants affected / at risk) | 59/138 | 58/138 | 339/692
Other Adverse Events (participants affected / at risk) | 133/138 | 133/138 | 643/692
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=138) | Arm B (Observation Only) (N=138) | All Participants (N=692)
Venous thrombosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vena cava thrombosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2)
Jugular vein thrombosis (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Surgical and medical procedures) | 0 (0) | 1 (1) | 3 (3)
Haemorrhagic vasculitis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Flushing (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peau D'orange (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 6 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 3 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 6 (6)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (4) | 5 (7)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Refractory Anaemia With An Excess Of Blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 4 (4)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nodal Marginal Zone B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Naevoid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 9 (9)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (3)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 7 (7)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 3 (4)
Complications of bone marrow transplant (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 8 (9)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 6 (6)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 18 (18)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 9 (9)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 14 (14) | 6 (7) | 54 (65)
Pneumocystis Jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pneumococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Perineal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Paraspinal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Myocarditis septic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myocarditis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 4 (4) | 7 (7)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6) | 10 (11)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (4)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 5 (5)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Immunosupression (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 4 (5)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 11 (16)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 5 (5)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2)
Infusion site erythema (General disorders) | 0 (0) | 1 (1) | 2 (5)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 5 (5)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 4 (4)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diverticular perporation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 10 (12)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Thyrotxic crisis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Cardic arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 7 (7)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic valve calcification (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (12) | 22 (29)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 36 (42)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 8 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A (N=138) | Arm B (Observation Only) (N=138) | All Participants (N=692)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 4 (4)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Spider vein (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 2 (3) | 6 (7)
Peripheral venous disease (Vascular disorders) | 3 (4) | 1 (1) | 4 (5)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 3 (3) | 19 (21)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 18 (27) | 5 (6) | 45 (57)
Hyperaemia (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 8 (16)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 1 (1) | 5 (5)
Flushing (Vascular disorders) | 2 (2) | 2 (2) | 8 (8)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0) | 2 (2)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 4 (6)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Nephrostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Mass excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
Cataract operation (Surgical and medical procedures) | 1 (1) | 4 (5) | 6 (8)
Astringent therapy (Surgical and medical procedures) | 1 (1) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (7) | 15 (20)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (6)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (8) | 19 (22)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 3 (5)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 8 (10)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 19 (24) | 18 (23) | 76 (97)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (14) | 9 (12) | 51 (61)
Prurigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (4) | 19 (22)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Hypertrichiosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 8 (8)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 15 (15)
Granulomatous rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 12 (14)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (7) | 29 (39)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 10 (11)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 1 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (7) | 23 (26)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 10 (11)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (3)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 14 (14)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 11 (11)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (5)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8) | 25 (28)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 6 (6)
Pharyngeal parasthesia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 5 (5) | 39 (40)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 8 (8)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4)
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 12 (15)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 11 (11) | 55 (62)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (4) | 14 (18)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (72) | 24 (37) | 135 (185)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 9 (10)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 7 (7)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 5 (6)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 2 (3)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 5 (5)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1) | 5 (5)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (3) | 5 (7)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Strangury (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 8 (9)
Renal cyst (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Renal atrophy (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 9 (10)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3) | 6 (6)
Nephroangiosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 5 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 6 (6) | 13 (14)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder hypertrophy (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Stress (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 5 (5)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8) | 5 (5) | 31 (33)
Feeling of despair (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 8 (8) | 2 (2) | 20 (20)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 9 (9) | 22 (23)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 3 (4) | 13 (15)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 2 (2) | 10 (10)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sensorimotor disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 4 (5) | 12 (14)
Presyncope (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 3 (3) | 10 (10)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 5 (5) | 9 (9) | 29 (29)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 8 (9) | 7 (8) | 23 (25)
Neuromuscular pain (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 2 (2) | 6 (6)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 4 (5)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 6 (8)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 16 (24) | 18 (25) | 68 (92)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Facial neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgraphia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (11) | 3 (3) | 17 (21)
Dysaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 16 (21) | 8 (8) | 36 (42)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 6 (6)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 7 (8)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 1 (3)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (3)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5) | 17 (19)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (11) | 43 (46)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 7 (8)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 14 (15)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 11 (12)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 16 (17)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 22 (22)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (7) | 25 (28)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 7 (8)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 3 (4)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (6)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 17 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 13 (19) | 62 (72)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (22) | 14 (23) | 52 (68)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Tetany (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 7 (9)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (10) | 1 (1) | 22 (31)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (7)
Hypoalbminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (9) | 3 (3) | 10 (13)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (5) | 2 (2) | 8 (11)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (6)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (6)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 7 (9) | 48 (56)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 11 (19) | 13 (21) | 46 (72)
Weight increased (Investigations) | 0 (0) | 1 (1) | 4 (6)
Weight decreased (Investigations) | 6 (7) | 4 (4) | 25 (27)
Transferrin saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (2) | 1 (1) | 5 (6)
Pulse abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Polymerase chain reaction positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 14 (20) | 10 (13) | 59 (96)
Oxygen saturation decrease (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 28 (65) | 29 (60) | 113 (289)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 13 (17) | 14 (23) | 45 (80)
Liver palpable (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Immunoglobulins decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Hypophonesis (Investigations) | 0 (0) | 0 (0) | 1 (1)
Histamine level increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 6 (8)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Coagulation time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 3 (3) | 3 (3)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2) | 17 (17)
Body temperature increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (3) | 1 (1) | 2 (4)
Blood pressure abnormal (Investigations) | 2 (2) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 1 (1) | 14 (16)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood immunoglobulin M decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 1 (1) | 0 (0) | 5 (5)
Blood glucose increased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Blood folate decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 4 (4) | 4 (5) | 12 (17)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 8 (9)
Biopsy prostate (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (4) | 11 (13)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (7) | 11 (20)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (4)
Tooth avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (3)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 5 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 23 (24)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 11 (12)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Dental restoration failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 6 (6)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Administration related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (3) | 1 (2) | 2 (5)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 7 (7)
Viral pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Viral parotitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 7 (8) | 2 (2) | 11 (12)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 2 (3) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 11 (14) | 14 (22) | 55 (73)
Ureaplasma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 24 (36) | 20 (26) | 63 (85)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 4 (4) | 1 (1) | 6 (6)
Tracheitis (Infections and infestations) | 3 (3) | 3 (3) | 8 (8)
Tooth infection (Infections and infestations) | 1 (2) | 2 (2) | 5 (6)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1) | 5 (5)
Tonsillitis (Infections and infestations) | 3 (3) | 2 (3) | 5 (6)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 2 (6) | 5 (9)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 14 (27) | 16 (21) | 45 (67)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 19 (21) | 9 (9) | 42 (46)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 3 (4)
Respiratory tract infection (Infections and infestations) | 4 (5) | 10 (19) | 24 (36)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Puncture site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Proteus infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (3)
Postoperative wound infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 17 (22) | 10 (13) | 44 (55)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (4) | 3 (6) | 9 (13)
Pertussis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 3 (6)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Oral infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 9 (17) | 4 (5) | 25 (35)
Oral fungal infection (Infections and infestations) | 2 (2) | 1 (2) | 5 (7)
Oral candidiasis (Infections and infestations) | 3 (3) | 3 (4) | 14 (15)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 2 (2) | 1 (2) | 4 (5)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 29 (55) | 24 (36) | 72 (120)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Nail infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1/1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 10 (15) | 5 (5) | 24 (32)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 17 (37) | 9 (14) | 46 (76)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
Labyrinthitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (3)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 20 (23) | 14 (18) | 56 (65)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 2 (3) | 0 (0) | 2 (3)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 16 (18) | 12 (12) | 46 (50)
Herpes virus infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (4)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hepatic infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 2 (3) | 2 (2) | 5 (6)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Gastrointestinal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 7 (7) | 11 (12)
Furuncle (Infections and infestations) | 1 (1) | 1 (4) | 4 (7)
Fungal skin infection (Infections and infestations) | 1 (2) | 2 (3) | 3 (5)
Fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 6 (6)
Folliculitis (Infections and infestations) | 1 (1) | 2 (5) | 8 (12)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Escherichia urinary tract infection (Infections and infestations) | 1 (2) | 2 (4) | 5 (8)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 3 (4) | 4 (4) | 14 (17)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Dacryocanaliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Cystitis Escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 4 (4) | 0 (0) | 6 (6)
Conjunctivitis (Infections and infestations) | 12 (14) | 4 (5) | 24 (27)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 8 (9)
Candida infection (Infections and infestations) | 3 (3) | 0 (0) | 5 (5)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Campylobacter colitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 24 (55) | 21 (27) | 78 (126)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Blastocystis infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bartholinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Balanitis candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Application site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Acute sinusitis (Infections and infestations) | 5 (6) | 1 (1) | 7 (7)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 4 (4)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Iodine allergy (Immune system disorders) | 1 (1) | 1 (1) | 2 (2)
Immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 9 (9) | 9 (9) | 26 (26)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 7 (7)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 5 (7)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 32 (45) | 29 (49) | 159 (258)
Puncture site pain (General disorders) | 1 (1) | 1 (1) | 3 (3)
Puncture site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Polyp (General disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 7 (8)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 3 (3) | 2 (2) | 8 (8)
Oedema peripheral (General disorders) | 6 (6) | 7 (8) | 38 (40)
Oedema (General disorders) | 3 (3) | 2 (2) | 9 (9)
Mucosal inflammation (General disorders) | 6 (6) | 7 (8) | 25 (27)
Malaise (General disorders) | 2 (2) | 1 (1) | 10 (10)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site thrombosis (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 3 (3)
Injection site reaction (General disorders) | 1 (2) | 1 (1) | 10 (13)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 8 (9)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site plaque (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 3 (3) | 6 (7) | 24 (34)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 0 (0) | 2 (3) | 2 (3)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 3 (3) | 8 (9)
Injection site induration (General disorders) | 3 (9) | 1 (2) | 5 (17)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 2 (2)
Injection site haematoma (General disorders) | 1 (2) | 0 (0) | 4 (5)
Injection site erythema (General disorders) | 10 (11) | 9 (14) | 38 (46)
Injection site discomfort (General disorders) | 2 (2) | 0 (0) | 2 (2)
Injection site discolouration (General disorders) | 1 (1) | 1 (1) | 3 (3)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 5 (5)
Infusion site rash (General disorders) | 0 (0) | 1 (1) | 2 (3)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion site inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 3 (3)
Infusion site erythema (General disorders) | 1 (6) | 0 (0) | 4 (16)
Influenza like illness (General disorders) | 6 (24) | 6 (9) | 20 (45)
Inflammation (General disorders) | 0 (0) | 1 (1) | 5 (6)
Implant site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 2 (2) | 0 (0) | 3 (7)
Hyperthermia (General disorders) | 3 (4) | 1 (1) | 7 (8)
Haemorrhagic cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 5 (5)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 4 (5)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 3 (3)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 30 (46) | 19 (25) | 115 (157)
Facial pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 1 (1) | 2 (2)
Chills (General disorders) | 8 (8) | 9 (9) | 40 (47)
Chest pain (General disorders) | 11 (12) | 7 (7) | 27 (29)
Chest discomfort (General disorders) | 3 (3) | 3 (3) | 10 (10)
Catheter site thrombosis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 27 (43) | 19 (28) | 113 (167)
Application site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Administration site inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Administration site extravasation (General disorders) | 1 (1) | 0 (0) | 3 (6)
Vomiting (Gastrointestinal disorders) | 23 (32) | 16 (31) | 96 (160)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 5 (5) | 2 (2) | 9 (9)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 3 (4) | 17 (18)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3) | 5 (5) | 15 (16)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (5) | 7 (10)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 45 (63) | 37 (65) | 199 (312)
Mouth ulceration (Gastrointestinal disorders) | 3 (4) | 3 (4) | 12 (15)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3) | 12 (12)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (13) | 7 (9) | 20 (24)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 12 (12)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (7)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 7 (7) | 26 (27)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 10 (10)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 35 (50) | 28 (36) | 143 (211)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 21 (26) | 15 (22) | 98 (129)
Colitis (Gastrointestinal disorders) | 3 (5) | 0 (0) | 6 (8)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Change in bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (6)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 11 (16) | 4 (5) | 39 (49)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 13 (15) | 13 (23) | 57 (74)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (8)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 2 (2) | 1 (1) | 6 (6)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 5 (5)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 3 (3)
Noninfective conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Eyelid swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1) | 2 (2) | 3 (3)
Eye pain (Eye disorders) | 4 (4) | 0 (0) | 6 (6)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Entropion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 0 (0) | 5 (5)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 2 (3) | 1 (2) | 5 (8)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 7 (10) | 2 (2) | 18 (21)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 2 (2) | 9 (10)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 2 (2) | 11 (12)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 3 (3)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Vantricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4) | 10 (10)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 4 (5) | 9 (11)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkinetic heart syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2) | 8 (12)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2) | 3 (4)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0) | 5 (5)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 4 (5) | 7 (8)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 10 (13) | 49 (75)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 48 (134) | 51 (173) | 226 (604)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (13) | 1 (1) | 16 (34)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 14 (47) | 9 (18) | 52 (126)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (8) | 15 (22)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 23 (35) | 21 (32) | 106 (172)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 2 (2) | 4 (5)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaldosteronism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (3)
Chloangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Choleithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 4 (6)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (3)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Porokeratosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 4 (4)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Spermatic cord mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Spermatic cord pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vascular operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT01461928/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT01461928/SAP_001.pdf